CLINICAL TRIAL: NCT05087134
Title: Characterizing Lymphangioleiomyomatosis (LAM) With 11C-Choline PET/CT
Brief Title: Characterizing LAM With 11C-Choline PET/CT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHLAM
Record Dates: First submitted 2021-09-14; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-09

CONDITIONS: Lymphangioleiomyomatosis
MeSH Terms: conditions — Lymphangioleiomyomatosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 11C-Choline PET/CT for Lymphangioleiomyomatosis (LAM) (Experimental): The patients were injected with 11C-Choline of 5-10mCi and underwent PET/CT scan 20~40min after the injection.
  Interventions: Drug: 11C-Choline

INTERVENTIONS:
Drug: 11C-Choline — 11C-Choline were injected into the patients before the PET/CT scans

SUMMARY:
It was reported that TSC2-deficient cells enhance phosphatidylcholine synthesis via the Kennedy pathway. 11C-Choline can reflect the metabolic process of choline in vivo by intravenous injection. The purpose of this study is the ability of 11C-Choline PET/CT to evaluate the baseline condition of LAM patients and the efficacy of rapamycin after treatment.

DETAILED DESCRIPTION:
Tuberous Sclerosis Complex (TSC) is an autosomal dominant disorder caused by inactivating mutations of the TSC1 or TSC2 gene, characterized by neurocognitive impairment and benign tumors of the brain, skin, heart, and kidneys. Lymphangioleiomyomatosis (LAM) is a diffuse proliferation of α-smooth muscle actin-positive cells associated with cystic destruction of the lung. LAM occurs almost exclusively in women, as a TSC manifestation or a sporadic disorder (TSC1/TSC2 somatic mutations). Biomarkers of whole-body tumor burden/activity and response to rapalogs or other therapies remain needed in TSC/LAM. It was reported that TSC2-deficient cells enhance phosphatidylcholine synthesis via the Kennedy pathway. 11C-Choline can reflect the metabolic process of choline in vivo by intravenous injection. The purpose of this study is the ability of 11C-Choline PET/CT to evaluate the baseline condition of LAM patients and the efficacy of rapamycin after treatment.

ELIGIBILITY:
Inclusion Criteria:

- provide a written informed consent; Diagnostic CT or MRI suggesting a diagnosis of lymphangioleiomyomatosis.

Exclusion Criteria:

- Females planning to bear a child recently or with childbearing potential; Known severe allergy or hypersensitivity to IV radiographic contrast； Inability to lie still for the entire imaging time.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value of 11C-Choline in LAM lesions | through study completion, an average of 2 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value (SUV) of the tracer in lymphatic lesion will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Li, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking union medical college hospital, Beijing, Dongcheng, China